CLINICAL TRIAL: NCT05755256
Title: Randomized, Double-blind, Placebo-controlled Trial to Assess the Impact of Probiotics on Skin Hydration in Adolescents and Young Adults with Mild Acne Vulgaris.
Brief Title: The Impact of Probiotics on Skin Hydration in Youth with Mild Acne
Acronym: YSH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lallemand Health Solutions (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: L-023
Record Dates: First submitted 2023-02-09; First posted 2023-03-06 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-07

CONDITIONS: Acne Vulgaris; Hydration Acne
Keywords: probiotics; acne; adolescents; young adults; skin hydration
MeSH Terms: conditions — Acne Vulgaris | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: This pilot study is a monocentric, randomized, double-blind, placebo-controlled, parallel-arm study. The product allocation will be performed using a dynamic randomization algorithm designed to minimize imbalance between the 2 arms, within the strata defined by 3 factors: age, Global Acne Evaluation (GEA) score and sex.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic (Experimental): The product contains the probiotic strain and no other ingredients.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): The control product is a placebo with the same characteristics of appearance and packaging as the tested product.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — After randomization, participants will consume the probiotic for 12 weeks.
  Arms: Probiotic
Dietary Supplement: Placebo — After randomization, participants will consume the placebo for 12 weeks.
  Arms: Placebo

SUMMARY:
The goal of this clinical trials is to test the impact of probiotics on skin hydration in adolescents and young adults with mild acne. The hypothesis of this study is that the probiotic formulation is superior to placebo in improving the skin hydration in adolescents and young adults with minimal acne after 12 weeks of consumption.

DETAILED DESCRIPTION:
This pilot study is a monocentric, randomized, double-blind, placebo-controlled, parallel-arm study. The product allocation will be performed using a dynamic randomization algorithm designed to minimize imbalance between the 2 arms, within the strata defined by 3 factors: age, Global Acne Evaluation (GEA) score and sex.

60 participants (adolescents and adults) with mild acne vulgaris will be recruited for this study, according to the following inclusion and exclusion criteria.

There will be a total of 3 study visits: V1 (screening and randomization), V2 (mid-study follow-up), and V3 (end-of-study). The study will last a total of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 15 and 26 years (limits included),
2. Suffering from mild acne vulgaris for at least 1 year (GEA score 1 or 2),
3. For women (adolescents and adults) who have started their sexual life: be menstruated and with the same reliable contraception method since at least six months before the beginning of the study and agreeing to keep it during the entire duration of the study. Following contraception methods are allowed: hormonal contraception, intra uterine device, surgical intervention, condoms with spermicides. Contraceptive implants (e.g. Nexplanon®) are not allowed. For women who have not started their sexual life yet, who do not intend to start their sexual life, who do not use a contraception: be menstruated and keep the habits unchanged;
4. For women (adolescents and adults): negative urine pregnancy test result;
5. Good general and mental health within the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or physical examination;
6. Agree to maintain the same skin care regimen throughout the study;
7. Able and willing to participate in the study by complying with the protocol procedures, as evidenced by their dated and signed informed consent form. For adolescents (15-17 years): informed consent form signed by the guardians/parents and the individual willing to participate;
8. Affiliated with a social security scheme. For adolescents: affiliated with the social security scheme of the guardians/parents;
9. Agreeing to be registered on the national file of volunteers in biomedical research file.

After 1 month following to the non-inclusion of the participant for failure to comply with one or more of the inclusion criteria listed above, a re-screening could be performed.

Exclusion Criteria:

1. GEA score <1 or > 2 (corresponding to the absence of acne or a moderate, severe or very severe acne vulgaris),
2. Any disease that affects the secretion of sex hormones,
3. Any other dermatological disease (psoriasis, atopic dermatitis, allergy, eczema, etc.);
4. Suffering from a metabolic disorder (diabetes, uncontrolled thyroidal condition, uncontrolled arterial hypertension, etc.) and/or from severe chronic disease (cancer, renal failure, HIV, immunodeficiency, hepatic or biliary disorders, arthritis, uncontrolled cardiac disease, etc.) or from a disease found to be inconsistent with the conduct of the study by the investigator;
5. Immunodeficiency (immunodeficient and immunocompromised participants, e.g. cancer, HIV, lymphoma, participants on long-term corticosteroid treatment, chemotherapy, and allograft participants);
6. Positive COVID-test results within the last 2 weeks and/or currently showing symptoms of COVID-19;
7. Use of any systemic antibiotic or oral zinc treatment within 4 weeks prior to randomization, or isotretinoin within 3 months prior to randomization.
8. Regular consumption of probiotics, fiber supplements, fermented milk, and/or yogurt containing probiotics within 2 weeks prior to randomization and agreeing not to consume this type of product during the whole study;
9. Use of hormone replacement therapy (including oral contraceptives) for less than 6 months;
10. Under treatment or dietary supplement which could significantly affect skin microbiota according to the investigator or stopped in a too short period before V1;
11. Use of topically applied products (including topical acne drug) that could modulate potential skin improvement within 4 weeks prior to randomization. This includes products with a pH ≥ 8 such as hormone treatments, retinoid and other skin cleansing products, Micellar waters pH ≤ 5 can be used without rubbing the skin too hard with a cotton wool pad in order not to induce a Köbner phenomenon (appearance of new acne lesions on healthy but traumatised skin);
12. UVA or UVB exposure in the last 4 weeks or expected exposure during the study (short daily sun exposure is acceptable). The use of a UVA and UVB protection sunscreen factor 50 is mandatory during the study to protect against UVs;
13. With a known or suspected food allergy or intolerance or hypersensitivity to ingredient of the study products (yeast);
14. Pregnant or lactating women or intending to become pregnant within 3 months ahead;
15. With significant change in dietary or physical activity habits in the 3 months before randomization and not agreeing to keep them unchanged throughout the study (hyper or hypocaloric diet, planned start or stop of sports activity in the next 3 months);
16. With a personal history of anorexia nervosa, bulimia, or significant eating disorders within 3 years prior to randomization;
17. Consuming more than 2 standard drinks daily of alcoholic beverages or not willing to maintain their drinking habits unchanged throughout the study;
18. Participating in another clinical trial or in the exclusion period of a previous clinical trial, or participating in cosmetic tests with or without patch tests or consumer tests with food supplements containing probiotics;
19. Smoking more than 5 cigarettes per day;
20. For adults (age ≥ 18 years): Under legal protection (guardianship, wardship) or deprived of his/her rights following an administrative or judicial decision;
21. Presenting psychological or linguistic incapability to sign the informed consent;
22. Impossible to contact in case of emergency;
23. Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros.

After 1 month following to the non-inclusion of the participant for failure to comply with one or more of the exclusion criteria listed above, a re-screening could be performed.

Ages: 15 Months to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Corneal hydration after 12 weeks | 12 weeks
  The primary endpoint of the study is to compare the absolute change of the hydration level of the facial cornea between baseline (visit V1) and visit V3, assessed with Corneometer® CM825 on the forehead expressed in arbitrary units (a.u.) ranging from 0 to 120 (<30: very dry skin; 30-40: dry skin; >40: normal hydrated skin).

SECONDARY OUTCOMES:
Corneal hydration of the forehead after 6 weeks | 6 weeks
  The absolute change of the hydration of the facial cornea measured on the forehead with Corneometer® CM825 (expressed in a.u.) between V1 and V2, ranging from 0 to 120 (<30: very dry skin; 30-40: dry skin; >40: normal hydrated skin)).
Transepidermal water loss of forehead skin | 12 weeks
  The absolute change of the transepidermal water loss (TEWL) measured on the forehead with Tewameter® TM300expressed in g/h/m² (0-10: very healthy; 10-15: healthy; 15-25: normal; 25-30: stretched skin; >30: critical), between V1 and each visit (V2, V3).
Symptoms of acne on face | 12 weeks
  The absolute change of acne vulgaris symptoms (face and back) assessed with the Échelle de Cotation des Lésions d'Acné (acne grading scale; ECLA) scale between V1 and each visit (V2, V3), expressed in a.u, ranging from 0 to 5 on the face (0: no lesions; 1: <5; 2: 5-9; 3: 10-19; 4: 20-40; 5: > 40 lesions), and ranging from 0 to 3 on the back (0: absent; 1: few; 2: moderate; 3: important).
Sebum levels on face | 12 weeks
  The absolute change of sebum level (expressed in μg/cm²) measured with Sebumeter® SM815 between V1 and V3, ranging from 0 to 350, on the forehead (<100: dry skin; 100-220: normal skin; >220: oily skin).
Disability caused by acne | 12 weeks
  The absolute change of disability caused by acne assessed with the Cardiff Acne Disability Index (CADI) score (expressed in a.u., range 0-15) between V1 and each visit (V2, V3).
Impact on quality of life | 12 weeks
  The absolute change of overall Quality of Life, general health and four quality of life domains (Physical, Psychological, Social Relationships and Environment) assessed with six sub-scores of the World Health Organization Quality of life questionnaire - Brief version (WHOQoL-BREF) (expressed in a.u., item scores range 1-5, transformed scores range 0-100) between V1 and each visit (V2, V3).
Self-assessment of acne level on face and back | 12 weeks
  The absolute change of self-assessment acne level assessed with a visual analogue scale (VAS, range 0-10) between V1 and each visit (V2, V3).
Self-assessment of treatment satisfaction | 12 weeks
  The global study product satisfaction assessed with a visual analogue scale VAS (range 0-10) at V2 and V3.

OTHER OUTCOMES:
Skin microbiota composition | 12 weeks
  The change in skin microbiota composition (by sequencing for V3-V4 regions of 16S rRNA genes) between V1 and V3. Comparisons will be made in terms of relative abundance at the Phylum, Family and Genus taxonomic ranks, alpha-diversity indices (observed richness, inverse Simpson and Shannon) and beta-diversity indices (Jaccard and Bray-Curtis).
Quantification of probiotic in stool samples | 12 weeks
  The change in the quantity of the probiotics (by qPCR) between V1 and V3 in stool samples.
Faecal microbiota composition | 12 weeks
  The change in fecal microbiota composition assessed via Shotgun metagenomic analysis at each visit V1, V2 and V3. Comparisons will be made in terms of relative abundance at the Phylum, Family, Genus and Species taxonomic ranks for bacterial and eukaryota compositions, alpha-diversity indices (observed richness, inverse Simpson and Shannon) and beta-diversity indices (Jaccard and Bray-Curtis).
Vital signs - heart rate | 12 weeks
  The absolute change in values between baseline (V1) and each visit (V2 and V3) for Heart Rate (HR, in bpm).
Vital signs - blood pressure | 12 weeks
  The absolute change in values between baseline (V1) and each visit (V2 and V3) for the Systolic Blood Pressure (SBP, in mmHg) and Diastolic Blood Pressure (DBP, in mmHg).
Frequency of adverse events | 12 weeks
  The frequency of adverse events (AEs): treatment emergent adverse events (TEAEs), treatment emergent serious adverse events (STEAEs), TEAEs leading to discontinuation of study product, treatment emergent adverse reactions (TEARs).
Gut tolerance of probiotic | 12 weeks
  The absolute change in values obtained with the Gastrointestinal Symptom Rating Scale (GSRS), which contains 15 items on a 7-point Likert scale (1 = "absence of troublesome symptoms", and 7 = "very troublesome symptoms"), between baseline (V1) and each visit (V2, V3).

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Metreau, M.D, Principal Investigator — BioFortis
Locations (1):
- Biofortis, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No
After publications of the results, de-identified data will be shared with qualified researchers and scientists upon reasonable request to the sponsor including a detailed proposal of the intended use of the data, as per the Lallemand Health Solutions Inc. Policy on Clinical Trial Transparency and Data Sharing (available upon request).